CLINICAL TRIAL: NCT03304301
Title: Effect of Sunlight Exposure and Outdoor Activities on Improving the Depression, Cognition and Quality of Life of the Institutionalized Elderly: A Randomized Controlled Trial
Brief Title: Effect of Sunlight Exposure and Outdoor Activities on Depression, Cognition and Quality of Life in the Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chiayi Christian Hospital (Other)
Collaborators: National Cheng Kung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 104114
Record Dates: First submitted 2017-10-02; First posted 2017-10-09 (Actual); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Aging; Nursing Homes; Depression in Old Age; Cognitive Impairment; Quality of Life
Keywords: sunlight exposure; institutionalized elderly; depression; quality of life; cognition function
MeSH Terms: conditions — Cognitive Dysfunction; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Participants will be encouraged to reduce time spent on bed and bedroom. We will also take participants outdoors and expose to sunlight (if the UV index is over 8 according to the forecast of Center Weather Bureau, the participants will be asked to stay inside) five days a week for three months.
  Interventions: Behavioral: sunlight exposure
- control group (No Intervention): Participants will receive routine care.

INTERVENTIONS:
Behavioral: sunlight exposure — Participants will be encouraged to reduce time spent on bed and bedroom. We will also take participants outdoors and receiving sunlight exposure (if the UV index is over 8 according to the forecast of Center Weather Bureau, the participants will be asked to stay inside) five days a week for three months
  Arms: experimental group

SUMMARY:
Background: The transition to long-term care facility can be a stressful and emotional event for the elderly. The evidences showed that the prevalence of depression and the cognition impairment were higher in the institutionalized elderly than the community dwelling elderly. It could affect the quality of life of the elderly and increase risk of mortality.

Purpose: The aim of the study is to evaluate the effect of outdoor activities and sunlight exposure on depression, cognitive function, and quality of life among institutionalized elderly.

Method: The design is a randomized control trial. Participants will be randomly allocated to experimental or control groups by block randomization. In the experimental group, participants will be encouraged to reduce time spent on bed and bedroom. Nurses, nurse aids or family will take participants outdoors and exposure their face, hands or arm to sunlight for 15-30 minutes a day, five days a week for three months (if the UV index is over 8 according to the forecast of Center Weather Bureau, the participants will be asked to stay inside). In the control group, the participants will receive routine care. The control group will neither be encouraged to stay outdoors nor limit the chance to exposure to sunlight.

Expected outcome: The expected benefit of the research is to improve the depression, cognitive function, and quality of life of the institutionalized elderly.

ELIGIBILITY:
Inclusion Criteria:

* resident in the long-term care facility for at least 6 months
* Barthel Index score is equal or over 20
* able to communicate
* life expectancy over 12 months
* conscious clear

Exclusion Criteria:

* allergy to sunlight
* diagnosed with skin cancer

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2016-06-30 (Actual); Primary Completion 2018-01-12 (Estimated); Study Completion 2018-04-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline depression at 3 months | baseline, three month after recruitment
  measured with GDS-15

SECONDARY OUTCOMES:
Change from baseline cognitive function at 3 months | baseline, three month after recruitment
  measured with SPMSQ

OTHER OUTCOMES:
Change from baseline quality of life at 3 months | baseline, three month after recruitment
  measured with EQ-5D

CONTACTS AND LOCATIONS:
Overall Officials: LIN TZUCHIA, MASTER, Principal Investigator — Chiayi christian hospital, Taiwan, R.O.C.
Locations (1):
- BaoKang Long-Term Care Center, Chiayi City, Taiwan

DOCUMENTS (1):
  • Study Protocol (2017-10-02): https://cdn.clinicaltrials.gov/large-docs/01/NCT03304301/Prot_000.pdf